CLINICAL TRIAL: NCT06557798
Title: Prospective, Multi-centre Clinical Investigation Evaluating the Outcomes of Patients Treated by Redo Transcatheter Aortic Valve Implantation for Bioprosthetic Valve Failure of a Transcatheter Aortic Valve
Brief Title: REdo Transcatheter Aortic VALVE Implantation for the Management of Transcatheter Aortic Valve Failure
Acronym: REVALVE
Status: Recruiting | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Collaborators: Medtronic (Industry); NAMSA (Other)
Responsible Party: Sponsor
Other Study IDs: CD23/157535
Record Dates: First submitted 2024-08-09; First posted 2024-08-16 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Aortic Valve Stenosis
Keywords: Bioprosthetic Valve Failure
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Redo TAVI: Redo Trans-catheter Aortic Valve Implantation for Bioprosthetic Valve Failure of a Trans-catheter Aortic Valve
  Interventions: Device: Any commercially available Edwards or Medtronic transcatheter aortic valve with the TAV-in-TAV (Redo TAVI) indication
- Explant: Surgical explantation with aortic valve replacement
  Interventions: Procedure: Surgical explantation and aortic valve replacement
- Optimal Medical Therapy: Conservative treatment, including optimal medical therapy +/- balloon aortic valvuloplasty
  Interventions: Other: Conservative management

INTERVENTIONS:
Device: Any commercially available Edwards or Medtronic transcatheter aortic valve with the TAV-in-TAV (Redo TAVI) indication — Redo TAVI will be performed using any commercially available Edwards or Medtronic transcatheter aortic valve platforms that have the TAV-in-TAV (Redo TAVI) indication according to the preferences of the local team in keeping with standard clinical care.
  Groups: Redo TAVI
Procedure: Surgical explantation and aortic valve replacement — Surgical explantation of all or part of the index transcatheter aortic valve, with open implantation of a new surgical or transcatheter aortic valve replacement will be performed according to the preferences of the local team in keeping with standard clinical care. Any commercially available approved surgical or transcatheter aortic valve may be used. Additional surgery, such as aortic root replacement, root enlargement, CABG, mitral valve repair/replacement, etc. will be performed at the discretion of the local team.
  Groups: Explant
Other: Conservative management — Conservative treatment, including optimal medical therapy +/- balloon aortic valvuloplasty
  Groups: Optimal Medical Therapy

SUMMARY:
Transcatheter aortic valve implantation (TAVI) is a key-hole technique to replace an aortic heart valve that is narrowed and/or leaking. Although TAVI is a safe and effective treatment for a faulty aortic heart valve, the new TAVI valve will not last forever. Because it is a 'tissue' valve (made from the lining of a cow or pig heart), the valve will fail after a period of time as the tissue degenerates.

When the TAVI valve fails, a viable treatment option is to perform a 'Redo TAVI' procedure, implanting a second TAVI valve inside the first failing valve.

The main purpose of this study is to carefully evaluate patients being treated by Redo TAVI in order to document the short-term and long-term outcomes of the procedure. The study will also obtain information about which factors predict those outcomes.

The study will also assess outcomes in patients who present with TAVI valve failure but are not suitable for Redo TAVI, and instead are treated either by open-heart surgery and surgical aortic valve replacement, or by medical therapy (medication).

The study will provide doctors the information they need to understand the best way to treat patients who present with TAVI valve failure, and in particular how to perform Redo TAVI procedures with the best possible outcomes for patients.

DETAILED DESCRIPTION:
To determine the acute and long-term outcomes of Redo Transcatheter Aortic Valve Implantation (TAVI) for the treatment of Bioprosthetic Valve Failure (BVF) affecting Transcatheter Aortic Heart Valves (THVs)

To determine the factors which predict the acute and long-term outcomes of Redo TAVI

To determine the proportion of patients presenting with BVF affecting THVs who are deemed unsuitable for Redo TAVI by the Heart Team

To determine the acute and long-term outcomes of surgical explantation and aortic valve replacement (AVR) for the treatment of BVF affecting THVs

To determine the survival of patients presenting with BVF affecting THVs who are managed conservatively - including optimal medical therapy (OMT) +/- balloon aortic valvuloplasty (BAV)

ELIGIBILITY:
Inclusion Criteria:

1. Bio-prosthetic Valve Failure (BVF) of a Transcatheter Aortic Valve requiring possible reintervention

Exclusion Criteria:

1. Bio-prosthetic Valve Failure due solely to paravalvular aortic regurgitation
2. Active endocarditis
3. Untreated acute valve thrombosis
4. Life-expectancy less than 1 year
5. Subject is less than legal age of consent, legally incompetent, or otherwise vulnerable
6. Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting to the Heart Team with bio-prosthetic valve failure affecting a transcatheter aortic valve
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2033-03 (Estimated)

PRIMARY OUTCOMES:
REVALVE success (Redo TAVI) | 30 days
  Correct positioning of a single prosthetic heart valve into the proper anatomic location, intended performance of the valve (mean gradient <20mmHg, peak velocity <3 m/s, Doppler velocity index ≥0.25. aortic regurgitation < moderate), Freedom from mortality, coronary obstruction, unplanned coronary revascularisation, surgery or intervention related to the device
Freedom from death/stroke/re-hospitalisation for valve or procedure-related causes (Redo TAVI) | 12 months
  Composite outcome of freedom from death/stroke/re-hospitalisation for valve or procedure-related causes
Valve Academic Research Consortium 3 (VARC3) Early Safety (EXPLANT) | 30 days
  Composite outcome of freedom from: death/stroke/VARC 3-4 bleeding/major vascular, access-related, or cardiac structural complication/AKI 3 or 4/moderate or severe AR/new permanent pacemaker/device-related surgery or intervention
Freedom from death/stroke/re-hospitalisation for valve or procedure-related causes (EXPLANT) | 12 months
  Composite outcome of freedom from death/stroke/re-hospitalisation for valve or procedure-related causes
Freedom from death/stroke/re-hospitalisation for valve or procedure-related causes (OMT) | 12 months
  Composite outcome of freedom from death/stroke/re-hospitalisation for valve or procedure-related causes

SECONDARY OUTCOMES:
Valve Academic Research Consortium 3 (VARC3) Technical Success (Redo TAVI and EXPLANT) | End of procedure
  Freedom from mortality, successful access, delivery of the device, and retrieval of the delivery system, correct positioning of a single prosthetic heart valve into the proper anatomical location, freedom from surgery or intervention related to the device or to a major vascular or access-related, or cardiac structural complication
Valve Academic Research Consortium 3 (VARC3) Device Success (Redo TAVI and EXPLANT) | 30 days
  Technical success, Freedom from mortality, Freedom from surgery or intervention related to the device, or to a major vascular or access-related or cardiac structural complication, Intended performance of the valve (mean gradient <20 mmHg, peak velocity <3 m/s, Doppler velocity index ≥0.25, aortic regurgitation < moderate)
Valve Academic Research Consortium 3 (VARC3) Early Safety (Redo TAVI) | 30 days
  Freedom from: death/stroke/VARC 2-4 bleeding (only VARC 3-4 for EXPLANT) /major vascular, access-related, or cardiac structural complication/Acute kidney injury (AKI) 3 or 4/moderate or severe Aortic Regurgitation/new permanent pacemaker/device-related surgery or intervention
Peak and mean invasive gradient post-procedure (Redo TAVI) | End of procedure
  Invasive pressure measurements
In-hospital Clinical Outcomes | Immediately after the procedure/surgery
  All-cause mortality; All stroke; Myocardial infarction; Coronary artery obstruction; Unplanned coronary revascularisation (PCI or CABG); Bleeding (VARC 1-4); Major or minor Vascular and access-related complications; Cardiac structural complications; Permanent pacemaker implantation; Acute kidney injury (AKI) stage 1-4; Endocarditis; Clinically significant valve thrombosis
Echocardiographic Assessment: Peak velocity | Pre-discharge or at 30 days, 1, 3, 5 years
  Peak velocity
Echocardiographic Assessment: Mean gradient | Pre-discharge or at 30 days, 1, 3, 5 years
  Mean gradient
Echocardiographic Assessment: Aortic valve area | Pre-discharge or at 30 days, 1, 3, 5 years
  Aortic valve area
Echocardiographic Assessment: Patient-prosthesis mismatch | Pre-discharge or at 30 days
  Patient-prosthesis mismatch
Echocardiographic Assessment: Aortic Regurgitation - paravalvular, transvalvular or total | Pre-discharge or at 30 days, 1, 3, 5 years
  Aortic Regurgitation - paravalvular, transvalvular or total
Echocardiographic Assessment: Left ventricular systolic function | Pre-discharge or at 30 days, 1, 3, 5 years
  Left ventricular systolic function
Clinical Outcomes | 1, 3 and 5 years
  All-cause mortality; Cardiovascular mortality; Valve-related mortality; Hospitalisation; Cardiovascular hospitalisation; Hospitalisation for valve or procedure-related causes; All stroke; Myocardial infarction; Coronary angiography; Coronary revascularization; Bioprosthetic valve dysfunction: i. Structural valve deterioration; ii. Non-structural valve deterioration (Prosthesis-patient mismatch, Paravalvular aortic regurgitation, Other) iii. Thrombosis iv. Endocarditis; Bioprosthetic valve failure; Aortic valve re-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Blackman, MD, Principal Investigator — Leeds Teaching Hospitals NHS Trust
Locations (53):
- Denmark (3):
  - Aalborg Universitethospital, Aalborg
  - Århus Universitetshospital, Aarhus
  - Rigshospitalet, Copenhagen
- Finland (2):
  - HUS Helsinki University Hospital, Helsinki
  - Turku University Hospital, Turku
- France (10):
  - Clinical Saint Augustin - Elsan, Bordeaux
  - Brest University Hospital Centre, Brest
  - Henri Mondor University Hospital, Créteil
  - ICPS Hôpital privé Jacques-Cartier, Massy
  - Hospital Marie Lannelongue, Paris
  - Institute Mutualiste Montsouris, Paris
  - Les Hospital Universitaires de Strasbourg, Strasbourg
  - Clinique Pasteur Toulouse, Toulouse
  - CHRU Hospitals of Tours, Tours
  - Medipole Lyon-Villeurbanne, Villeurbanne
- Germany (9):
  - Kerckhoff Klinik, Bad Nauheim
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Klinikum Dortmund GmbH - St. Johannes Hospital, Dortmund
  - Herzzentrum Dresden Universitätsklinik, Dresden
  - Universitatsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Schleswig-Holstein (UKSH), Kiel
  - HELIOS Herzzentrum Leipzig GmbH, Leipzig
  - Universitätsklinikum Schleswig-Holstein (UKSH), Lübeck
  - LMU Klinikum, München
- Shaare Zedek Medical Center, Jerusalem, Israel
- Italy (4):
  - Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele, Catania
  - Centro Cardiologico Monzino, Milan
  - IRCSS Policlinico San Donato, San Donato Milanese
  - Ospedale Borgo Trento - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Netherlands (3):
  - Amphia Hospital, Breda
  - Maastricht University Medical Center (MUMC), Maastricht
  - Erasmus University Medical Center, Rotterdam
- Norway (2):
  - Haukeland Sykehus, Bergen
  - Oslo University Hospital, Oslo
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Skånes Universitetssjukhus Lund, Lund
  - Nya Karolinska Sjukhuset Solna, Solna
- Switzerland (2):
  - Inselspital - Universitätsspital Bern, Bern
  - Luzerner Kantonsspital, Lucerne
- United Kingdom (14):
  - Queen Elizabeth Hospital, Birmingham
  - Royal Sussex County Hospital, Brighton
  - Bristol Royal Infirmary, Bristol
  - University Hospital of Wales, Cardiff
  - Golden Jubilee National Hospital, Glasgow
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Glenfield Hospital, Leicester
  - Guys and St Thomas' NHS Foundation Trust, London
  - St. George's Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Popma JJ, Deeb GM, Yakubov SJ, Mumtaz M, Gada H, O'Hair D, Bajwa T, Heiser JC, Merhi W, Kleiman NS, Askew J, Sorajja P, Rovin J, Chetcuti SJ, Adams DH, Teirstein PS, Zorn GL 3rd, Forrest JK, Tchetche D, Resar J, Walton A, Piazza N, Ramlawi B, Robinson N, Petrossian G, Gleason TG, Oh JK, Boulware MJ, Qiao H, Mugglin AS, Reardon MJ; Evolut Low Risk Trial Investigators. Transcatheter Aortic-Valve Replacement with a Self-Expanding Valve in Low-Risk Patients. N Engl J Med. 2019 May 2;380(18):1706-1715. doi: 10.1056/NEJMoa1816885. Epub 2019 Mar 16. PMID 30883053
- [Background] Mack MJ, Leon MB, Thourani VH, Makkar R, Kodali SK, Russo M, Kapadia SR, Malaisrie SC, Cohen DJ, Pibarot P, Leipsic J, Hahn RT, Blanke P, Williams MR, McCabe JM, Brown DL, Babaliaros V, Goldman S, Szeto WY, Genereux P, Pershad A, Pocock SJ, Alu MC, Webb JG, Smith CR; PARTNER 3 Investigators. Transcatheter Aortic-Valve Replacement with a Balloon-Expandable Valve in Low-Risk Patients. N Engl J Med. 2019 May 2;380(18):1695-1705. doi: 10.1056/NEJMoa1814052. Epub 2019 Mar 16. PMID 30883058
- [Background] Vahanian A, Beyersdorf F, Praz F, Milojevic M, Baldus S, Bauersachs J, Capodanno D, Conradi L, De Bonis M, De Paulis R, Delgado V, Freemantle N, Gilard M, Haugaa KH, Jeppsson A, Juni P, Pierard L, Prendergast BD, Sadaba JR, Tribouilloy C, Wojakowski W; ESC/EACTS Scientific Document Group. 2021 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2022 Feb 12;43(7):561-632. doi: 10.1093/eurheartj/ehab395. No abstract available. PMID 34453165
- [Background] Otto CM, Nishimura RA, Bonow RO, Carabello BA, Erwin JP 3rd, Gentile F, Jneid H, Krieger EV, Mack M, McLeod C, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A, Toly C. 2020 ACC/AHA Guideline for the Management of Patients With Valvular Heart Disease: Executive Summary: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2021 Feb 2;143(5):e35-e71. doi: 10.1161/CIR.0000000000000932. Epub 2020 Dec 17. PMID 33332149
- [Background] Fukuhara S, Brescia AA, Deeb GM. Surgical Explantation of Transcatheter Aortic Bioprostheses: An Analysis From the Society of Thoracic Surgeons Database. Circulation. 2020 Dec 8;142(23):2285-2287. doi: 10.1161/CIRCULATIONAHA.120.050499. Epub 2020 Dec 7. No abstract available. PMID 33284653
- [Background] Bapat VN, Zaid S, Fukuhara S, Saha S, Vitanova K, Kiefer P, Squiers JJ, Voisine P, Pirelli L, von Ballmoos MW, Chu MWA, Rodes-Cabau J, DiMaio JM, Borger MA, Lange R, Hagl C, Denti P, Modine T, Kaneko T, Tang GHL; EXPLANT-TAVR Investigators. Surgical Explantation After TAVR Failure: Mid-Term Outcomes From the EXPLANT-TAVR International Registry. JACC Cardiovasc Interv. 2021 Sep 27;14(18):1978-1991. doi: 10.1016/j.jcin.2021.07.015. PMID 34556271
- [Background] Tuzcu EM, Kapadia SR, Vemulapalli S, Carroll JD, Holmes DR Jr, Mack MJ, Thourani VH, Grover FL, Brennan JM, Suri RM, Dai D, Svensson LG. Transcatheter Aortic Valve Replacement of Failed Surgically Implanted Bioprostheses: The STS/ACC Registry. J Am Coll Cardiol. 2018 Jul 24;72(4):370-382. doi: 10.1016/j.jacc.2018.04.074. PMID 30025572
- [Background] Testa L, Agnifili M, Van Mieghem NM, Tchetche D, Asgar AW, De Backer O, Latib A, Reimers B, Stefanini G, Trani C, Colombo A, Giannini F, Bartorelli A, Wojakowski W, Dabrowski M, Jagielak D, Banning AP, Kharbanda R, Moreno R, Schofer J, van Royen N, Pinto D, Serra A, Segev A, Giordano A, Brambilla N, Popolo Rubbio A, Casenghi M, Oreglia J, De Marco F, Tanja R, McCabe JM, Abizaid A, Voskuil M, Teles R, Biondi Zoccai G, Bianchi G, Sondergaard L, Bedogni F. Transcatheter Aortic Valve Replacement for Degenerated Transcatheter Aortic Valves: The TRANSIT International Project. Circ Cardiovasc Interv. 2021 Jun;14(6):e010440. doi: 10.1161/CIRCINTERVENTIONS.120.010440. Epub 2021 Jun 7. PMID 34092097
- [Background] Landes U, Sathananthan J, Witberg G, De Backer O, Sondergaard L, Abdel-Wahab M, Holzhey D, Kim WK, Hamm C, Buzzatti N, Montorfano M, Ludwig S, Conradi L, Seiffert M, Guerrero M, El Sabbagh A, Rodes-Cabau J, Guimaraes L, Codner P, Okuno T, Pilgrim T, Fiorina C, Colombo A, Mangieri A, Eltchaninoff H, Nombela-Franco L, Van Wiechen MPH, Van Mieghem NM, Tchetche D, Schoels WH, Kullmer M, Tamburino C, Sinning JM, Al-Kassou B, Perlman GY, Danenberg H, Ielasi A, Fraccaro C, Tarantini G, De Marco F, Redwood SR, Lisko JC, Babaliaros VC, Laine M, Nerla R, Castriota F, Finkelstein A, Loewenstein I, Eitan A, Jaffe R, Ruile P, Neumann FJ, Piazza N, Alosaimi H, Sievert H, Sievert K, Russo M, Andreas M, Bunc M, Latib A, Godfrey R, Hildick-Smith D, Chuang MA, Blanke P, Leipsic J, Wood DA, Nazif TM, Kodali S, Barbanti M, Kornowski R, Leon MB, Webb JG. Transcatheter Replacement of Transcatheter Versus Surgically Implanted Aortic Valve Bioprostheses. J Am Coll Cardiol. 2021 Jan 5;77(1):1-14. doi: 10.1016/j.jacc.2020.10.053. PMID 33413929
- [Background] Forrestal BJ, Case BC, Yerasi C, Shea C, Torguson R, Zhang C, Ben-Dor I, Deksissa T, Ali S, Satler LF, Shults C, Weissman G, Wang JC, Khan JM, Waksman R, Rogers T. Risk of Coronary Obstruction and Feasibility of Coronary Access After Repeat Transcatheter Aortic Valve Replacement With the Self-Expanding Evolut Valve: A Computed Tomography Simulation Study. Circ Cardiovasc Interv. 2020 Dec;13(12):e009496. doi: 10.1161/CIRCINTERVENTIONS.120.009496. Epub 2020 Dec 4. PMID 33272031
- [Background] Ochiai T, Oakley L, Sekhon N, Komatsu I, Flint N, Kaewkes D, Yoon SH, Raschpichler M, Patel V, Tiwana R, Enta Y, Mahani S, Kim Y, Stegic J, Chakravarty T, Nakamura M, Cheng W, Makkar R. Risk of Coronary Obstruction Due to Sinus Sequestration in Redo Transcatheter Aortic Valve Replacement. JACC Cardiovasc Interv. 2020 Nov 23;13(22):2617-2627. doi: 10.1016/j.jcin.2020.09.022. PMID 33213747
- [Background] Landes U, Richter I, Danenberg H, Kornowski R, Sathananthan J, De Backer O, Sondergaard L, Abdel-Wahab M, Yoon SH, Makkar RR, Thiele H, Kim WK, Hamm C, Buzzatti N, Montorfano M, Ludwig S, Schofer N, Voigtlaender L, Guerrero M, El Sabbagh A, Rodes-Cabau J, Mesnier J, Okuno T, Pilgrim T, Fiorina C, Colombo A, Mangieri A, Eltchaninoff H, Nombela-Franco L, Van Wiechen MPH, Van Mieghem NM, Tchetche D, Schoels WH, Kullmer M, Barbanti M, Tamburino C, Sinning JM, Al-Kassou B, Perlman GY, Ielasi A, Fraccaro C, Tarantini G, De Marco F, Witberg G, Redwood SR, Lisko JC, Babaliaros VC, Laine M, Nerla R, Finkelstein A, Eitan A, Jaffe R, Ruile P, Neumann FJ, Piazza N, Sievert H, Sievert K, Russo M, Andreas M, Bunc M, Latib A, Bruoha S, Godfrey R, Hildick-Smith D, Barbash I, Segev A, Maurovich-Horvat P, Szilveszter B, Spargias K, Aravadinos D, Nazif TM, Leon MB, Webb JG. Outcomes of Redo Transcatheter Aortic Valve Replacement According to the Initial and Subsequent Valve Type. JACC Cardiovasc Interv. 2022 Aug 8;15(15):1543-1554. doi: 10.1016/j.jcin.2022.05.016. Epub 2022 Jul 13. PMID 35926921
- [Background] Carroll JD, Mack MJ, Vemulapalli S, Herrmann HC, Gleason TG, Hanzel G, Deeb GM, Thourani VH, Cohen DJ, Desai N, Kirtane AJ, Fitzgerald S, Michaels J, Krohn C, Masoudi FA, Brindis RG, Bavaria JE. STS-ACC TVT Registry of Transcatheter Aortic Valve Replacement. Ann Thorac Surg. 2021 Feb;111(2):701-722. doi: 10.1016/j.athoracsur.2020.09.002. Epub 2020 Nov 16. PMID 33213826
- [Derived] Blackman DJ, Aktaa S, Pickles D, Abdel-Wahab M, De Backer O, Van Mieghem NM, Treede H, Landes U, Bapat V, Hildick-Smith D, Barbanti M. REdo transcatheter aortic VALVE implantation for the management of transcatheter aortic valve failure: Design and rationale of the REVALVE study. Int J Cardiol. 2025 Sep 15;435:133400. doi: 10.1016/j.ijcard.2025.133400. Epub 2025 May 18. PMID 40393632